CLINICAL TRIAL: NCT01185873
Title: The Effect of Hepatic Impairment on the Pharmacokinetics of RO5190591/Ritonavir: A Multiple-Center, Open-Label Study Following Multiple Oral Doses of RO5190591/Ritonavir to Subjects With Mild, Moderate, or Severe Hepatic Impairment and Healthy Subjects With Normal Hepatic Function
Brief Title: A Study of Danoprevir in Healthy Volunteers And Patients With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP25290; 2010-020314-29
Record Dates: First submitted 2010-08-17; First posted 2010-08-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danoprevir; Ritonavir

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: danoprevir; Drug: ritonavir

INTERVENTIONS:
Drug: danoprevir — Repeated oral doses
Drug: ritonavir — Repeated oral doses

SUMMARY:
This non-randomized, multi-center, open-label study will evaluate the pharmacokinetics and the safety and tolerability of danoprevir (RO5190591) and ritonavir in healthy volunteers and patients with mild, moderate or severe hepatic impairment. Participants will be administered repeated daily doses of danoprevir and ritonavir. The anticipated time on study treatment is 10 days.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

* Adult healthy volunteers, 18-70 years of age
* Weight >/=50.0 kg
* Body Mass Index (BMI) 18.0-40.0 kg/m2
* Ability and willingness to abstain from alcohol-containing beverages or food from 48 hours prior to entry in the clinical study center until discharge
* Ability and willingness to abstain from grapefruit or grapefruit juice, star fruit, and Seville oranges from 7 days prior to entry in the clinical study center until discharge
* Medical history without major recent or ongoing pathology

Patients with hepatic impairment:

* Adult patients, 18-70 years of age
* Weight >/=50.0 kg
* Body Mass Index (BMI) 18.0-40.0 kg/m2
* Ability and willingness to abstain from alcohol-containing beverages or food from 48 hours prior to entry in the clinical study center until discharge
* Ability and willingness to abstain from grapefruit or grapefruit juice, star fruit, and Seville oranges from 7 days prior to entry in the clinical study center until discharge
* Stable, mild, moderate, or severe liver disease of cryptogenic, post-hepatic, hepatitis B or alcoholic origin

Exclusion Criteria:

Healthy Volunteers:

* Pregnant or lactating women and male partners of women who are pregnant or lactating
* Uncontrolled treated/untreated hypertension (systolic blood pressure >/=160 mmHg and /or diastolic blood pressure >/=105 mmHg
* Any history of clinically significant cardiovascular or cerebrovascular disease
* Creatinine clearance </=60 mL/min
* Positive test results for drugs or alcohol
* Donation or loss of blood over 450 ml within 60 days prior to screening

Patients with hepatic impairment:

* Pregnant or lactating women and male partners of women who are pregnant or lactating
* Uncontrolled treated/untreated hypertension (systolic blood pressure >/=160 mmHg and /or diastolic blood pressure >/=105 mmHg
* Any history of clinically significant cardiovascular or cerebrovascular disease
* Severe ascites at screening or admission to the clinic
* History of or current severe hepatic encephalopathy (grade 3 or higher)
* Any evidence of progressive liver disease within the last 4 weeks
* History of liver transplantation
* Creatinine clearance </=60 mL/min
* Positive test results for drugs or alcohol
* Donation or loss of blood over 450 ml within 60 days prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (plasma concentration) of danoprevir in patients with hepatic impairment | From baseline to day 10

SECONDARY OUTCOMES:
Safety and tolerability (incidence of adverse events) of danoprevir in patients with hepatic impairment | From baseline to day 10

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Lenexa, Kansas, United States
- Prague, Czechia
- Bratislava, Slovakia